CLINICAL TRIAL: NCT00174980
Title: An Open Label, Proof of Concept Study, to Evaluate the Safety and Biological Effects of Oxycyte™ Perfluorocarbon in Patients With A Severe Head Injury Requiring Intracranial Pressure Monitoring-OX-CL-II-002
Brief Title: Study of Oxycyte in Severe Closed Head Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tenax Therapeutics, Inc. (Industry)
Collaborators: Virginia Commonwealth University (Other)
Responsible Party: Timothy Bradshaw, SVP Clinical Development, Oxygen Biotherapeutics, Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OX-CL-II-002
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2008-10

CONDITIONS: Traumatic Brain Injury
Keywords: Oxycyte; perfluorocarbon oxygen carrier; brain oxygen tension
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — perfluoro(t-butylcyclohexane)

INTERVENTIONS:
Drug: perfluorocarbon emulsion (Oxycyte) infusion — one time dose of 3mL/kg over 15 minutes
  Other Names: Oxycyte

SUMMARY:
Brain damage as a result of decreased oxygen to the brain is found in 80% of patients that die with severe head injuries. Laboratory studies in animals and clinical trials have shown that increasing oxygen in the brain results in better brain oxygen consumption, less cell death, and better functional outcome. This study will test the hypothesis that Oxycyte is an effective way to increase brain oxygen levels in severe head injury.

DETAILED DESCRIPTION:
Decreased brain oxygen in severe brain injuries appears to be implicated in poor functional outcome and death. Animal and clinical studies have shown that increasing brain oxygen in such patients improves functional outcome, and Oxycyte has been shown to be an effective means of delivering oxygen to tissues, including the brain. This study is an eight patient proof of concept study to test the effects of oxygen delivery with Oxycyte in patients with a severe traumatic head injury with a Glasgow Coma Scale (GCS) score of 3 to 9.

Subjects diagnosed with a severe head injury (GCS 3-9) who receive a brain oxygen monitor and microdialysis catheter, will undergo baseline monitoring for 4 hours. In the first 4 subjects the Fi02 on the ventilator will be increased to 50% for a 4 hour stabilization period and this will be followed by a single intravenous infusion of 3ml/kg of Oxycyte. The Fi02 will remain at 50% for 24 hours.

In the second 4 subjects the Fi02 on the ventilator will be increased to 100% for a 4 hour stabilization period and this will be followed by a single intravenous infusion of 3ml/kg of Oxycyte. The Fi02 will remain at 100% for 24 hours.

Subjects will be enrolled, treated, and then monitored by LICOX 02 monitor before and after infusion of PFC, and then for at least 48 hours following the discontinuation of Oxycyte.

ELIGIBILITY:
Inclusion Criteria:

* severe closed head injury patients or GCS 3-9 patients who receive brain oxygen monitoring
* ventriculostomy/ICP monitor
* at least one reactive pupil
* no known life threatening disease prior to trauma
* age 18-70 years old
* consent for microdialysis/brain 02 monitoring
* legal family representative present that can give informed consent for perfluorocarbon administration

Exclusion Criteria:

* no motor response
* both pupils fixed and dilated
* no consent available
* allergy to egg proteins
* coagulopathy
* major liver injury
* major pulmonary injury

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2005-09; Primary Completion 2008-01 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Increase in Brain Oxygen Tension levels in severe traumatic head injury patients with GCS score of 3-9

SECONDARY OUTCOMES:
Adverse events will be captured throughout drug infusion and 2 weeks post, Severe adverse events will be captured for 6 months. Glascow outcomes score at 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: M. R Bullock, M.D., Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University Medical Center, Richmond, Virginia, United States